CLINICAL TRIAL: NCT00493155
Title: "An Open-label, Multiple Ascending Dose Study to Determine the Maximum Tolerated Dose of R1530 in Patients With Advanced Solid Tumors."
Brief Title: A Multiple Ascending Dose Study of R1530 in Patients With Advanced Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NO18674
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RG1530

INTERVENTIONS:
Drug: RG1530 — Administered po at escalating doses (10 cohorts)

SUMMARY:
This study will determine the maximum tolerated dose, and assess the safety, tolerability and pharmacokinetics of R1530 administered orally to patients with advanced or metastatic solid tumors. R1530 will be administered daily for 14 days at the starting dose; this dose will be escalated in subsequent cohorts of patients, after a satisfactory assessment of safety and tolerability of the previous dose, until the maximum tolerated dose is reached. The anticipated time on study treatment is until disease progression, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* cancer not amenable to curative treatment (ie advanced and/or metastatic);
* measurable or evaluable disease;
* adequate cardiac, hepatic and renal function.

Exclusion Criteria:

* patients with known CNS metastases;
* serious cardiovascular illness or other medical conditions;
* prior chemotherapy, radiotherapy or immunotherapy within 28 days of start of treatment , or hormone therapy within 14 days of start of treatment;
* inability to swallow oral medications, or impaired gastrointestinal absorption.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | Throughout study

SECONDARY OUTCOMES:
AEs, laboratory parameters | Throughout study
Plasma levels of R1530 | Throughout study
Tumor assessments | Every 2 cycles of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- United States (4):
  - Boston, Massachusetts
  - Detroit, Michigan
  - Las Vegas, Nevada
  - Houston, Texas